CLINICAL TRIAL: NCT00178425
Title: Pharmacokinetics of Intravenous / Oral MMF and Oral Tacrolimus in Live Donor and Deceased Donor Liver Transplant Patients
Brief Title: PK of MMF in Cadaveric vs Living Donor Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSRB 10410; CEL 458
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Transplantation, Liver
Keywords: mycophenolate mofetil hydrochloride; pharmacokinetics; tacrolimus
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Serial blood sampling as described in protocol
Procedure: Estimation of Creatinine Clearance at regular intervals

SUMMARY:
The purpose of this study is to measure the amount of MMF and tacrolimus concentration in the blood at a given time. Currently MMF is ordered as a set dose and tacrolimus is given based on body weight. While the deceased donor transplant receives the complete liver, in the live donor just over half of the liver is given (about 60%). The way these different types of transplants break down drugs could be different. Measuring the drug levels allows us to know what happens to the medication in between the morning and the evening dose.

DETAILED DESCRIPTION:
The purpose of this study is to measure the amount of MMF and tacrolimus concentration in the blood at a given time. Currently MMF is ordered as a set dose and tacrolimus is given based on body weight. While the deceased donor transplant receives the complete liver, in the live donor just over half of the liver is given (about 60%). The way these different types of transplants break down drugs could be different. Measuring the drug levels allows us to know what happens to the medication in between the morning and the evening dose.

12 subjects with live liver donors and 12 subjects with deceased donors will be included in the study.

Each patient will have 12 (twelve) blood samples (half a teaspoon) drawn at 0,1, 2, 3, 4, 4½; 5, 6, 7, 8, 10 and 12 hours from an intravenous line placed during the operation. At the same time, 24-hour urine will be collected to measure your kidney function. After 4 to 6 days post transplant when the will be switched to oral MMF, again 10 (ten) blood samples a half teaspoon each will be drawn at 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours. Blood will be drawn with the routine daily blood work for the first 14 days and then at 1 and 3 months after transplant. Total blood drawn over 3 months will be about 7 tablespoons. A 24-hour urine will be collected in a container given to you starting one day before the routine clinic visit (as a standard of care). The 24-hour urine will be collected at 1 and 3 months after transplant as well.

If a woman, who could become pregnant, a pregnancy test will be done before your transplant. They would also have to use birth control during the study period and 6 months after the completion of study.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Female patients
* Negative pregnancy test
* Willing for contraception during the study period and 6 weeks after study

Exclusion Criteria:

* Serum Creatinine > 2.5 mg/dl
* On Dialysis
* HIV +ve
* Re-transplantation
* On Ventilator
* Multi-organ Transplant
* Platelets < 50,000
* WBC < 2,500

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Comparison of Pharmacokinetics of MMF in living donor liver transplant and deceased donor liver transplant

SECONDARY OUTCOMES:
Comparison of Pharmacokinetics of IV MMF vs PO MMF
Pharmacokinetics of tacrolimus after liver transplant

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Jain, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States